CLINICAL TRIAL: NCT01683916
Title: Chonnam National University Hospital IRB
Brief Title: Anesthetic Requirement and Stress Hormone Response During Surgery in Spinal Cord-injured Patients
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Kyung Yeon Yoo, Professor, Chonnam National University Hospital
Other Study IDs: 2010-12-198
Record Dates: First submitted 2012-09-08; First posted 2012-09-12 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2010-12

CONDITIONS: Complete Spinal Cord Injury; Surgery
Keywords: spinal cord injury; stress hormone; surgery; bispectral index value; volatile anesthetic
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Spinal cord injury (SCI) reduces anesthetic requirements and stress hormonal responses. Anesthetic requirements and stress hormone response are compared in SCI patients undergoing anesthesia with sevoflurane supplemented with clinically equivalent doses of either N2O or remifentanil.

DETAILED DESCRIPTION:
Nitrous oxide (N2O) is often used for anesthetic adjuvant, but may be associated with side effects and toxicities. Remifentanil shares characteristics with N2O, including anesthetic-reducing and antinociceptive effects and a rapid recovery. Anesthetic requirements and stress hormone response in SCI patients undergoing anesthesia with sevoflurane supplemented with clinically equivalent doses of either N2O or remifentanil. Forty-five SCI patients scheduled to undergo pressor sore surgery below the level of the injury are randomly allocated to receive either sevoflurane alone (control, n=15), or combined with 67% N2O (n=15) or target-controlled infusions of 1.37 ng/mL remifentanil (n=15). Sevoflurane concentration is titrated to maintain a Bispectral Index (BIS) value of 40-50. Measurements include end-tidal sevoflurane concentrations, mean arterial blood pressure (MAP), heart rate (HR), and plasma catecholamine and cortisol concentrations.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II, with chronic, clinically complete cord injuries scheduled for a surgery for pressure sore below the level of the neurologic lesion under general anesthesia.

Exclusion Criteria:

* Cardiovascular, pulmonary, or metabolic diseases. Patients who took medications that would influence autonomic or cardiovascular responses to the surgery

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ASA physical status II, with chronic, clinically complete cord injuries scheduled for a surgery for pressure sore below the level of the neurologic lesion under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Gwangju, South Korea